CLINICAL TRIAL: NCT05688943
Title: Comparative Analysis of Spinal Versus General Anesthesia for Vaginal Natural Orifice Transluminal Endoscopic Tubal Sterilization: A Prospective, Randomized Controlled Trial
Brief Title: Comparative Analysis of Spinal Anesthesia Versus General Anesthesia for vNOTES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Meredith Gray, Associate Professor, Obstetrics & Gynecology, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00149365
Record Dates: First submitted 2022-12-14; First posted 2023-01-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Tubal Ligation
Keywords: vNOTES; Tubal Sterilization; Regional Anesthesia; laparoscopy
MeSH Terms: interventions — Anesthesia, Spinal; Anesthesia, Conduction; Anesthesia, General; Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: This a a randomized control trail that will have 2 groups. One will be the control group and will receive the standard of care, general anesthesia. The other group will be the experimental group which will receive spinal anesthesia in place in general anesthesia.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): This arm will receive general anesthesia for vNOTES surgery.
  Interventions: Procedure: General Anesthesia
- Spinal Anesthesia (Experimental): This arm will receive spinal anesthesia for vNOTES surgery.
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: Spinal Anesthesia — Fentanyl (1µg/kg) and midazolam are administered intravenously prior to puncture. Using an aseptic technique, the subarachnoid space is punctured with a 25/27 gauge needle in the intervertebral space, and a standard dose of chloroprocaine 45-60mg is injected. Alternative spinal anesthetics include bupivacaine 6-15mg and mepivacaine 50-70mg. The participant is then placed in the supine position in 10-degree Trendelenburg until the lack of sensitivity is adequate at spinal level T4.
  Other Names: Regional Anesthesia
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — General anesthesia is a state of controlled unconsciousness. During a general anesthetic, medicines are used to send the participant to sleep making the participant unaware of surgery and so that the participant does not move or feel pain while the surgery is carried out. Induction of general anesthesia includes the use intravenous sedative-hypnotic agents such as propofol, etomidate, or ketamine, along with adjuvant agents such as fentanyl, lidocaine, or midazolam. A neuromuscular blocking agent such as succinylcholine or rocuronium is used to facilitate endotracheal intubation.
  Other Names: Endotracheal intubation
  Arms: General Anesthesia

SUMMARY:
This study compares general anesthesia and spinal anesthesia for vNOTE tubal sterilization. A direct comparison of these methods has not been done before for this surgical approach. Investigators will aim to compare the two methods to determine the differences in perioperative complications, postoperative pain, postoperative nausea and vomiting, and the time to get the patient ready for discharge from the recovery room.

DETAILED DESCRIPTION:
Anesthesia is a controlled, temporary loss of sensation or awareness used to perform surgical procedures. Spinal anesthesia is commonly used in obstetrics and gynecology for vaginal procedures as well as cesarean sections. The use of spinal anesthesia for laparoscopic surgery is an adequate and safe alternative to general anesthesia which remains the gold standard. Vaginal Natural Orifice Endoscopic Surgery (vNOTES) is a minimally invasive laparoscopic approach used for tubal sterilization that is currently performed under general anesthesia. This study is proposing that spinal anesthesia is an adequate and safe alternative to general anesthesia for vNOTES tubal sterilization. If participants join the study, all other routine care will continue but the researchers will randomly assign participants, like flipping a coin, to one of two groups. Both types of anesthesia are commonly used but the researchers are doing this study because it is not known if spinal anesthesia is a better alternative than general anesthesia which is typically used. The goal is to find out what might be best for future patients. If it turns out the two types of anesthesia are about the same, then surgeons would know that choosing the type with fewer side effects still gives satisfactory results and allows for this surgery to be performed safely. The risks involved in participating in this study are the same as all other anesthetic and surgical procedures which have significant physical risks. If participants choose to enroll, there will be a 50/50 chance of being assigned to either the standard of care group which will receive general anesthesia or the experimental group which will receive spinal anesthesia. Benefits cannot be guaranteed but, It is possible participants could be assigned to a type of anesthesia that has fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21years old keeping in line with regulations posed by federally funded insurance programs
* cis-female or gender non-conforming person with female reproductive organs
* request for permanent sterilization
* no prior hysterectomy or trachelectomy
* undergoing tubal sterilization only or salpingo-oophorectomy only for cancer risk reduction due to genetic pre-disposition
* non-emergent/scheduled outpatient procedure
* non-pregnant, ≥6 weeks postpartum
* American Society of Anesthesia (ASA) physical status classification I or II
* All subjects must be determined to be appropriate candidates for VNOTES by the surgeon based on the review of medical and surgical history
* Those undergoing additional procedures such as insertion or removal of a long-acting reversible contraceptive (Intrauterine device or subdermal implant) may be included.

Exclusion Criteria:

* Ectopic pregnancy, ovarian torsion, or adnexal mass requiring urgent or emergent treatment;
* Trans-masculine person considering surgical masculinization due to additional surgeries involved;
* Undergoing adnexal surgery for suspected or confirmed malignancy;
* History of endometriosis, or other inflammatory diseases that have been determined to add to the complexity and increase the risk of injury with vaginal surgery;
* prior genital surgery or congenital abnormality that would prevent vaginal access;
* prior spinal surgery or severe scoliosis that would hinder placement and effective functioning of neuraxial anesthetics;
* uncorrected thrombocytopenia or coagulopathy;
* ASA physical status classification ≥III.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis-female or gender non-conforming person
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative complications performing VNOTES tubal sterilization with Spinal Anesthesia | during surgery
  This study seeks to explore the feasibility of performing vaginal natural orifice transluminal endoscopic surgery (VNOTES) tubal sterilization under small-dose spinal anesthesia compared to the gold standard, general anesthesia, in healthy patients and to analyze intraoperative complications.
Incidence of perioperative complications performing VNOTES tubal sterilization with Spinal Anesthesia | up to 7 days after surgery
  This study seeks to explore the feasibility of performing vaginal natural orifice transluminal endoscopic surgery (VNOTES) tubal sterilization under small-dose spinal anesthesia compared to the gold standard, general anesthesia, in healthy patients and to analyze postoperative complications.

SECONDARY OUTCOMES:
Rate of post-operative pain between patients | immediately after the surgery
  To determine the differences in postoperative pain between patients in each anesthesia group based on a pain scale assessed post-operatively.
Occurrence of postoperative nausea/vomiting | immediately after the surgery
  To determine the differences in the occurrence of postoperative nausea/vomiting (PONV) in a yes or no survey question.
Compare time until PACU discharge-to-home readiness between patients | immediately after the surgery
  To determine the differences in time until post-anesthesia care unit (PACU) discharge-to-home readiness between patients postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith K Gray, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States